CLINICAL TRIAL: NCT01675128
Title: A Phase I/II Study of ISIS 183750 in Combination With Irinotecan in Irinotecan-refractory Colorectal Cancer
Brief Title: ISIS 183750 With Irinotecan for Advanced Solid Tumors or Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Tim Greten, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120187; 12-C-0187
Record Dates: First submitted 2012-08-25; First posted 2012-08-29 (Estimated); Results first posted 2016-04-25 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-03

CONDITIONS: Colorectal Neoplasms; Colorectal Carcinoma; Colorectal Tumors
Keywords: Human Eukaryotic Translation Initiation Factor 4E (eIF4E) protein; Refractory; Oncogene; Maximum Tolerated Dose; Safety
MeSH Terms: conditions — Colorectal Neoplasms | interventions — LY 2275796; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Phase I Dose Level I (Experimental): Irinotecan 160 mg/m^2 every other week; ISIS 183750 started 800 mg/every week will be administered intravenously on Cycle 1 Days 1, 3, 5, 8, 15 and 22 of a 28 day cycle, restaged every 8 weeks.
  Interventions: Drug: ISIS 183750; Drug: Irinotecan
- Phase I Dose Level II (Experimental): Irinotecan 180 mg/m^2 every other week; ISIS 183750 1000 mg/every week will be administered intravenously on Cycle 1 Days 1, 3, 5, 8, 15 and 22 of a 28 day cycle, restaged every 8 weeks.
  Interventions: Drug: ISIS 183750; Drug: Irinotecan
- Phase II Dose Level I (Experimental): Irinotecan 160 mg/m^2 every other week; ISIS 183750 1000mg every week will be administered as an intravenous infusion every week without break, i.e. Days 1, 8, 15 and 22 of a 28-day cycle. Patients will be re-staged every 8 weeks.
  Interventions: Drug: ISIS 183750; Drug: Irinotecan

INTERVENTIONS:
Drug: ISIS 183750
Drug: Irinotecan

SUMMARY:
Background:

- Irinotecan is a drug that is used to treat colon or rectal cancer. It affects the deoxyribonucleic acid (DNA) of growing cancer cells. It is most often used with other chemotherapy drugs. Researchers want to test it with an experimental drug, ISIS 183750. They want to see if the drugs are a safe and effective treatment for advanced solid tumors or colorectal cancer that has not responded to other treatments.

Objectives:

- To test the safety and effectiveness of ISIS 183750 with irinotecan for advanced solid tumors or colorectal cancer.

Eligibility:

- Individuals at least 18 years of age who have solid tumors or colorectal cancer that has not responded to other treatments.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will also be collected. Tumor tissue samples may be collected as well before and after treatment. Imaging studies will also be performed.
* Participants will take ISIS 183750 once a week for 28-day cycles of treatment. On the first cycle, they will also have ISIS 183750 on days 3 and 5.
* Participants will take irinotecan every second week, beginning on day 15 of the first cycle.
* Treatment will be monitored with frequent blood tests and imaging studies.
* Treatment will continue as long as the cancer does not grow and the side effects are not severe.

DETAILED DESCRIPTION:
Background:

The eukaryotic translation initiation factor - eIF4E - is a potent oncogene that is found to be dysregulated in approximately 30% of human cancers. Upregulation of eIF4E is an early event in colorectal cancer (CRC) and correlates with CRC progression. ISIS 183750 is a second-generation antisense oligonucleotide (ASO) designed to inhibit the production of the human eukaryotic translation initiation factor 4E (eIF4E) protein.

Objectives:

Primary:

To establish Maximum Tolerated Dose (MTD) and establish safety for the combination of ISIS 183750 and irinotecan in advanced solid tumors.

Secondary:

* To evaluate Response Rate, Progression Free Survival (PFS), Overall Survival (OS) for the combination of ISIS 183750 and irinotecan in advanced irinotecan-refractory colorectal cancer.
* To perform correlative studies to evaluate the effect of eIF4E inhibition on relevant regulated proteins and immune cells.
* To characterize the plasma pharmacokinetic (PK) parameters for ISIS 183750 in the absence and presence of irinotecan
* To characterize the plasma PK parameters for irinotecan in the presence of ISIS 183750

Eligibility:

-Adult patients with irinotecan-resistant colorectal cancer (or advanced solid tumor in phase I part).

Design:

* This is a single-arm phase I/II study whereby all patients will receive the combination of ISIS 183750 and irinotecan. All cycles are 28 days.
* Cycle 1 only: ISIS 183750 will be administered intravenously on Cycle 1 Days 1, 3, 5, 8, 15 and 22.
* Cycle 2 and beyond: ISIS 183750 will be administered as an intravenous infusion every week without break, i.e. Days 1, 8, 15 and 22 of a 28-day cycle. Patients will be re-staged every 8 weeks.
* Irinotecan will be administered at a dose of 160mg/m^2 as an intravenous infusion every second week commencing on Day 15 of Cycle 1. The primary endpoint of the study will be to establish maximum tolerated dose (MTD) for the combination of ISIS 183750 and irinotecan in advanced solid tumors. The phase II portion of the study will be confined to irinotecan-refractory colorectal cancer. Irinotecan-refractory will be defined as patients who have radiological evidence of disease progression whilst receiving irinotecan or within 3 months after completing it.
* Correlative studies will comprise: Mandatory pre- and post- dose biopsies for eIF4e messenger ribonucleic acid (mRNA) and protein (IHC) analysis will be performed in the phase II portion of the study; Immune subsets; positron emission tomography (PET) responses (only in expansion cohort); Pharmacokinetic data regarding the interaction of irinotecan and ISIS183750 in 10-12 patients.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Phase I: Patients must have histopathological confirmation of carcinoma by the Laboratory of Pathology of the National Cancer Institute (NCI) prior to entering this study.
* Phase II: Patients must have histopathological confirmation of Colorectal Carcinoma (CRC) by the Laboratory of Pathology of the NCI prior to entering this study. For this portion of the study patients must also have irinotecan-refractory colorectal cancer and have also received prior treatment for advanced/metastatic disease with an oxaliplatin-, bevacizumab-, or epidermal growth factor receptor (EGFR) inhibitor-containing (only for subjects with wild type Kras) regimen. Irinotecan-refractory will be defined as patients who have radiological evidence of disease progression whilst receiving irinotecan or within 3 months after completing it.
* Patients must have disease that is not amenable to potentially curative resection or ablative techniques and have received at least one prior standard chemotherapeutic regimen for metastatic disease.
* All patients enrolled will be required to have measurable disease. For the phase II portion of the study patients must have disease that is amenable to biopsy and be willing to undergo this.
* Age greater than18 years
* Life expectancy of greater than 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Patients must have acceptable organ and marrow function as defined below:

  * leukocytes > 3,000/mcL
  * absolute neutrophil count > 1,500/mcL
  * platelets > 100,000/mcL
  * total bilirubin Within normal institutional limits
  * Serum albumin greater than or equal to 2.5 g/dL
  * Patients are eligible with alanine aminotransferase (ALT) or aspartate aminotransferase (AST) measuring 3 x upper limit of normal (ULN) if no liver metastasis or up to 5 x ULN with liver metastasis.
  * creatinine < 1.5X institution upper limit of normal
  * OR
  * creatinine clearance > 45 mL/min/1.73 m^2, as calculated below, for patients with creatinine levels above institutional normal
  * Estimated creatinine clearance (mL/min)

    * Females see calculations
    * Males see calculations - May use a 24 hr. urine collection to determine creatinine clearance.
  * Measured creatinine clearance (mL/min)
* Patients must have recovered from any acute toxicity related to prior therapy, including surgery. Toxicity should be < grade 1 or returned to baseline.
* Patients must not have other invasive malignancies within the past 3 years (with the exception of non-melanoma skin cancers, carcinoma in situ of the cervix and noninvasive bladder cancer that has had successful curative treatment).
* The effects of ISIS 183750 on the developing human fetus are unknown. For this reason women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 3 months after dosing with study medication ceases. However, adequate contraception for male patients should be used for 16 weeks post- last dose due to sperm life cycle. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Women of child-bearing potential must have a negative pregnancy test prior to entry.
* Patient must be able to understand and willing to sign a written informed consent document.
* Men and women of all races and ethnic groups are eligible for this trial.
* Ejection fraction > 55% on echocardiogram.

EXCLUSION CRITERIA:

* Patients who have had chemotherapy (or so-called targeted systemic therapy), large field radiotherapy, or major surgery must wait 4 weeks after completing treatment prior to entering the study.
* Patients may not be receiving any antineoplastics or other drugs intended to treat cancer within 4 weeks prior to starting ISIS 183750.
* Patients with known brain metastases will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Patients with clinically significant ascites, pleural effusion, and/or peripheral edema, unless the ascites or pleural effusion occurred as a result of malignancy.
* Patients with known hypersensitivity to irinotecan.
* Patients with known homozygous mutations in the UTG1A1 UUDP-glucuronosyltransferase 1-1) allele, or with unknown UTG1A1 status but who could not tolerate irinotecan even after dose reduction.
* Patients with bleeding diathesis and subjects who are receiving anticoagulation treatment with International Normalized Ratio (INR) > 2.5 are excluded.
* Uncontrolled intercurrent illness including, but not limited to, hypertension (systolic blood pressure (BP) > 160, diastolic BP > 100), ongoing or active systemic infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia or psychiatric illness/social situations that would limit compliance with study requirements.
* Human immunodeficiency virus (HIV)-positive patients receiving anti-retroviral therapy are excluded from this study due to the possibility of pharmacokinetic interactions between antiretroviral medications and the investigational agent.
* Known hepatitis B or hepatitis C infection.
* Pregnancy and breast feeding are exclusion factors. Enrolled patients must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, the duration of study participation and 3 months after the end of the treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-08; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim F Greten, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Result] Duffy AG, Makarova-Rusher OV, Ulahannan SV, Rahma OE, Fioravanti S, Walker M, Abdullah S, Raffeld M, Anderson V, Abi-Jaoudeh N, Levy E, Wood BJ, Lee S, Tomita Y, Trepel JB, Steinberg SM, Revenko AS, MacLeod AR, Peer CJ, Figg WD, Greten TF. Modulation of tumor eIF4E by antisense inhibition: A phase I/II translational clinical trial of ISIS 183750-an antisense oligonucleotide against eIF4E-in combination with irinotecan in solid tumors and irinotecan-refractory colorectal cancer. Int J Cancer. 2016 Oct 1;139(7):1648-57. doi: 10.1002/ijc.30199. Epub 2016 Jun 27. PMID 27194579
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-C-0187.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I Dose Level II: Irinotecan 180 mg/m^2 every other week; ISIS 183750 1000mg every week will be administered intravenously on Cycle 1 Days 1, 3, 5, 8, 15 and 22 of a 28 day cycle, restaged every 8 weeks.
Period: Overall Study
Arm/Group | Phase I Dose Level I | Phase I Dose Level II | Phase II Dose Level I
Started | 4 | 10 | 10
Completed | 2 | 8 | 9
Not Completed | 2 | 2 | 1
Not completed — Disease progression on study | 1 | 1 | 1
Not completed — Refused further treatment | 1 | 0 | 0
Not completed — Pulmonary complication; off study | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase I Dose Level I: Irinotecan 160 mg/m^2 every other week; ISIS 183750 started 800mg/every week will be administered intravenously on Cycle 1 Days 1, 3, 5, 8, 15 and 22 of a 28 day cycle, restaged every 8 weeks.
- Phase I Dose Level II: Irinotecan 180 mg/m^2 every other week; ISIS 183750 1000mg/every week will be administered intravenously on Cycle 1 Days 1, 3, 5, 8, 15 and 22 of a 28 day cycle, restaged every 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Phase I Dose Level I | Phase I Dose Level II | Phase II Dose Level I | Total
Number analyzed (Participants) | 4 | 10 | 10 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 5 | 7 | 15
  >=65 years | 1 | 5 | 3 | 9
Age, Continuous [Median (Full Range); unit: years] | 61.6 [54.7 to 73.15] | 65.7 [43.37 to 79.64] | 60.6 [50.4 to 72.7] | 62.7 [43.4 to 79.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 4 | 10
  Male | 2 | 6 | 6 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 10 | 10 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 2 | 6
  White | 3 | 7 | 7 | 17
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 10 | 10 | 24

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of ISIS 183750 in Advanced Solid Tumors
Description: MTD is the dose level at which no more than 1 of up to 6 patients experience dose-limiting toxicity (DLT) during the first 6 weeks of treatment, and no dose below that which at least 2 (of </=6) patients have DLT as a result of the drug.
Time Frame: 2 years
Measure: Number; unit: mg
Groups:
- All Phase I Participants: ISIS 183750 started 800mg/every week will be administered intravenously on Cycle 1 Days 1, 3, 5, 8, 15 and 22 of a 28 day cycle, restaged every 8 weeks.
Arm/Group | All Phase I Participants
Number analyzed (Participants) | 14
mg | 1000

2. Primary Outcome: Maximum Tolerated Dose of Irinotecan in Advanced Solid Tumors
Description: as for outcome 1
Time Frame: 2 years
Measure: Number; unit: mg/m^2
Groups:
- All Phase I Participants: Irinotecan 160 (and 180) mg/m^2 every other week.
Arm/Group | All Phase I Participants
Number analyzed (Participants) | 14
mg/m^2 | 160

3. Primary Outcome: Number of Participants With a Change in the Level of a Particular Gene Called elF4E [Eukaryotic Initiation Factors (elF)4e Messenger Ribonucleic Acid (mRNA) Levels] in Matched Pre and Post Tumor Biopsies
Description: A change in elF4e levels is defined as an increase or decrease compared to baseline and is measured between two time points before rand after 2 weeks of treatment by quantitative real-time reverse transcription polymerase chain reaction (qRT-PCR).
Time Frame: 2 weeks
Population: Mandatory pre- and post-dose biopsies for elF4e messenger ribonucleic acid (mRNA) analysis was performed in the phase II portion of the study.
Measure: Number; unit: participants
Groups:
- Phase II Dose Level I: Irinotecan 160 mg/m^2 every other week; ISIS 183750 1000mg/every week will be administered as an intravenous infusion every week without break, i.e. Days 1, 8, 15 and 22 of a 28-day cycle. Patients will be re-staged every 8 weeks.
Arm/Group | Phase II Dose Level I
Number analyzed (Participants) | 9
participants | 5

4. Primary Outcome: Number of Participants With a Change in elF4e Protein Levels in Matched Pre and Post Tumor Biopsies
Description: A change in protein is defined as an increase or decrease compared to baseline and is measured between two time points by immunohistochemistry (IHC) analysis.
Time Frame: 2 weeks
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Phase II Dose Level I
Number analyzed (Participants) | 9
participants | 5

5. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: 21 months
Measure: Number; unit: participants
Arm/Group | Phase I Dose Level I | Phase I Dose Level II | Phase II Dose Level I
Number analyzed (Participants) | 4 | 10 | 10
participants | 4 | 10 | 10

6. Secondary Outcome: Objective Response
Description: Objective response was evaluated by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete Response (CR) is the disappearance of all target lesions. Any pathological lymph nodes (whether target or non target) must have reduction in short axis to <10mm. Partial response (PR) is at least a 30% reduction in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Progressive disease (PD) is at least a 20% increase in the sum of athe diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more lesions is also considered progression).
Time Frame: up to 2 cycles
Population: Only 6/10 participants in Phase I, Dose Level II and 9/10 participants in Phase II were evaluable for response. Per protocol, no responses were to be reported for the Phase I Dose Level I Arm because the participants have different histologies, thus there are no objective responses for Phase I Dose Level I.
Measure: Number; unit: participants
Groups:
- Phase I Dose Level 2: Irinotecan 180 mg/m^2 every other week; ISIS 183750 1000mg/every week will be administered intravenously on Cycle 1 Days 1, 3, 5, 8, 15 and 22 of a 28 day cycle, restaged every 8 weeks.
Arm/Group | Phase I Dose Level 2 | Phase II Dose Level I
Number analyzed (Participants) | 6 | 9
participants
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 0 | 0
  Stable Disease (SD) | 3 | 4
  Progressive (PD) | 3 | 5

7. Secondary Outcome: Number of Participants With Progression Free Survival
Description: Progression free survival is defined as the time beginning on the on study date and continuing until date of progression or date removed from study for an adverse event.
Time Frame: ≤ 6 months
Population: Only 6/10 participants in Phase I, Dose Level II and 9/10 participants in Phase II were evaluable. Per protocol, progression free survival was not to be reported for the Phase I Dose Level I Arm because the participants have different histologies, thus there is no progression free survival data for Phase I Dose Level I.
Measure: Number; unit: participants
Arm/Group | Phase I Dose Level II | Phase II Dose Level I
Number analyzed (Participants) | 6 | 9
participants | 3 | 6

8. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from the on study date until the date of death or date last known alive.
Time Frame: ≥ 12 months
Population: Only 6/10 participants in Phase I, Dose Level II and 9/10 participants in Phase II were evaluable. Per protocol, overall survival was not to be reported for the Phase I Dose Level I Arm because the participants have different histologies, thus overall survival data for Phase I Dose Level I.
Measure: Number; unit: participants
Arm/Group | Phase I Dose Level II | Phase II Dose Level I
Number analyzed (Participants) | 6 | 9
participants | 1 | 1

9. Secondary Outcome: AUC(ALL) (Area Under the Plasma Concentration vs. Time Curve for All Time Points)
Description: AUC(ALL) (Area under the plasma concentration vs. time curve for all time points) was assessed for CPT-11 (irinotecan), its active metabolite SN38, and the glucuronic acid metabolite of SN38, SN38-G to derive the total AUC(ALL).
Time Frame: up to 24 hours post end of infusion
Population: Phase I Dose Level I and Phase I Dose Level II were grouped together for this outcome measure. Complete pharmacokinetic data for only ten of the fourteen participants enrolled on the phase I portion of the study were available for analysis. Data is unavailable to report each individual time point.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Groups:
- Phase I Dose Level I & Phase I Dose Level II: Irinotecan 160 mg/m^2 every other week; ISIS 183750 started 800 mg/every week will be administered intravenously on Cycle 1 Days 1, 3, 5, 8, 15 and 22 of a 28 day cycle, restaged every 8 weeks.
  Phase I Dose Level II Irinotecan 180 mg/m^2 every other week; ISIS 183750 1000mg/every week will be administered intravenously on Cycle 1 Days 1, 3, 5, 8, 15 and 22 of a 28 day cycle, restaged every 8 weeks.
Arm/Group | Phase I Dose Level I & Phase I Dose Level II
Number analyzed (Participants) | 10
hr*ng/mL
  CPT-11 (irinotecan) | 9016 (1793)
  SN38 | 119 (42.3)
  SN38-G | 1340 (751)

10. Secondary Outcome: Number of Participants With Intracellular and Stromal Presence of ISIS in Tumor Tissue
Description: Intracellular and stromal presence of ISIS in tumor tissue was assessed by immunohistochemistry (IHC) and Crystal Violet staining to determine effectiveness of drug. Tissue that retains stain indicates intracellular and stromal presence of ISIS and determines if the drug is working. Relative staining intensity (intensity criteria unavailable) was evaluated by a pathologist.
Time Frame: 2 weeks
Population: Per protocol, this outcome measure was assessed in the phase II portion only because all participants were getting the same dose.
Measure: Number; unit: participants
Arm/Group | Phase II Dose Level I
Number analyzed (Participants) | 10
participants | 10

11. Secondary Outcome: Number of Participants With a Reduced Effect of elF4E Inhibition on Relevant Regulated Proteins
Description: Protein levels in the biopsy sample was assessed by immunohistochemistry using anti-oligonucleotide antibody to assess the downstream effect and determine if proteins are being manufactured. The number of participants with a reduced effect (criteria unavailable) of elF4E inhibition on relevant regulated proteins determines if the drug is working.
Time Frame: 2 weeks
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Phase II Dose Level I
Number analyzed (Participants) | 10
participants | 10

12. Secondary Outcome: Number of Participants With a Decrease in elF4E mRNA Expression in Peripheral Blood
Description: Peripheral blood analysis of elF4E mRNA expression was performed using real time quantitative polymerase chain reaction (q-PCR) to assess the downstream effect and determine if proteins are being manufactured. The number of participants with a decrease (criteria unavailable) in elF4E determines if the drug is working. Cell proliferation or reduction was evaluated by a pathologist.
Time Frame: 2 weeks
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Phase II Dose Level I
Number analyzed (Participants) | 10
participants | 10

ADVERSE EVENTS:
Arm/Group | Phase I Dose Level I | Phase I Dose Level II | Phase II Dose Level I
Serious Adverse Events (participants affected / at risk) | 3/4 | 3/10 | 4/10
Other Adverse Events (participants affected / at risk) | 4/4 | 10/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Dose Level I (N=4) | Phase I Dose Level II (N=10) | Phase II Dose Level I (N=10)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 | 1 (1) | 1 (1)
Confusion (Psychiatric disorders) | 0 | 0 | 1 (1)
Creatinine increased (Investigations) | 0 | 0 | 1 (1)
Death Not otherwise specified (NOS) (General disorders) | 2 (2) | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 2 (2)
Dysarthria (Nervous system disorders) | 0 | 0 | 1 (1)
Fatigue (General disorders) | 0 | 0 | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1)
Hematoma (Vascular disorders) | 0 | 0 | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 (1)
Hypotension (Vascular disorders) | 0 | 1 (1) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 | 1 (1)
Neutrophil count decreased (Investigations) | 0 | 1 (1) | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 (1) | 0
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 | 0
Serum amylase increased (Investigations) | 1 (1) | 0 | 0
Thromboembolic event (Vascular disorders) | 1 (1) | 1 (1) | 0
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1 (1) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Dose Level I (N=4) | Phase I Dose Level II (N=10) | Phase II Dose Level I (N=10)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 4 (7) | 7 (23) | 7 (14)
Agitation (Psychiatric disorders) | 0 | 0 | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 6 (19) | 8 (31)
Alkaline phosphatase increased (Investigations) | 2 (3) | 6 (14) | 9 (24)
Allergic reaction (Immune system disorders) | 0 | 0 | 1 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 4 (13) | 8 (28) | 9 (26)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 5 (8) | 5 (7)
Anxiety (Psychiatric disorders) | 0 | 0 | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 6 (10) | 7 (18)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 | 1 (1)
Blood bilirubin increased (Investigations) | 0 | 1 (1) | 3 (4)
Blurred vision (Eye disorders) | 0 | 0 | 1 (1)
Chills (General disorders) | 0 | 2 (2) | 2 (3)
Confusion (Psychiatric disorders) | 1 (1) | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 3 (3) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0
Creatinine increased (Investigations) | 1 (2) | 3 (21) | 4 (9)
Dehydration (Metabolism and nutrition disorders) | 0 | 3 (3) | 4 (6)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0
Diarrhea (Gastrointestinal disorders) | 3 (6) | 6 (14) | 9 (17)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 | 0
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0
Edema limbs (General disorders) | 1 (1) | 3 (4) | 3 (5)
Edema trunk (General disorders) | 0 | 0 | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1)
Eye pain (Eye disorders) | 0 | 0 | 1 (1)
Fatigue (General disorders) | 3 (5) | 4 (7) | 7 (10)
Fever (General disorders) | 0 | 6 (8) | 7 (12)
Flu like symptoms (General disorders) | 0 | 2 (2) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1)
Headache (Nervous system disorders) | 0 | 1 (1) | 6 (6)
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 2 (5) | 3 (8)
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 (1) | 1 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1 (2) | 1 (2)
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1 (2) | 1 (2)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 2 (4) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (10) | 9 (36) | 9 (35)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 1 (3) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 (8) | 5 (11) | 3 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2) | 1 (4) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (4) | 4 (5) | 9 (20)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (3) | 6 (11) | 6 (14)
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 2 (2)
Infusion related reaction (General disorders) | 0 | 1 (2) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 0 | 2 (2)
Lymphocyte count decreased (Investigations) | 4 (22) | 6 (27) | 0
Malaise (General disorders) | 1 (1) | 0 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 6 (11) | 6 (10)
Neutrophil count decreased (Investigations) | 3 (9) | 6 (35) | 4 (7)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 (1)
Pain (General disorders) | 1 (1) | 2 (2) | 6 (10)
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 3 (5) | 7 (25) | 6 (11)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1)
Presyncope (Nervous system disorders) | 0 | 0 | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 (2) | 2 (2)
Serum amylase increased (Investigations) | 0 | 0 | 1 (2)
Sinusitis (Infections and infestations) | 0 | 0 | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4) | 4 (5) | 4 (4)
Weight loss (Investigations) | 2 (2) | 3 (3) | 2 (2)
White blood cell decreased (Investigations) | 4 (18) | 8 (51) | 7 (17)
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1)
Edema face (General disorders) | 0 | 2 (3) | 0
Hematuria (Renal and urinary disorders) | 0 | 1 (1) | 0
Bloating (Gastrointestinal disorders) | 0 | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 | 1 (1) | 1 (1)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 (2) | 1 (2)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 0 | 2 (2) | 2 (2)
Paresthesia (Nervous system disorders) | 0 | 1 (1) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1 (2) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3 (3) | 3 (3)
Rectal pain (Gastrointestinal disorders) | 0 | 1 (1) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1 (1) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 | 1 (1) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 (1) | 1 (1)
Nervous system disorders- Other, specify (alteration in smell) (Nervous system disorders) | 0 | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No